CLINICAL TRIAL: NCT05421208
Title: Cardiovascular Autonomic and Immune Mechanism of Post COVID-19 Tachycardia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 220763; 967054 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Post-acute COVID-19 Syndrome; Postural Tachycardia Syndrome (POTS); Long COVID; SARS CoV 2 Infection
Keywords: SARS-CoV-2 infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Case-control study
Who Masked: Participant
Masking Description: The POTS patients will be randomized to chronic transcutaneous vagus nerve stimulation (tVNS) in any of the two sites on ear, and there will 50% change to be allocated to one of the sites that may have less stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Compare inflammatory markers (IL-6) in post- COVID 19 POTS patients with Controls (Experimental): Biochemical endpoints: Measurement of Inflammatory markers (especially IL-6) in both Post- COVID-19 POTS patients and compare it with controls.
  Controls are the participants who recovered from COVID 19 infection with no sequelae
  Interventions: Diagnostic Test: Levels of inflammatory cytokine ( IL-6) in post-COVID-19 POTS and controls; Diagnostic Test: Levels of inflammatory cytokine ( IL-6) in controls
- Effect of OI symptoms & inflmmation after Restoring PNS functions in post-COVID POTS patients. (Experimental): Effects of restoring PNS function in post-COVID-19 POTS patients with chronic transcutaneous vagus nerve stimulation (tVNS) on inflammation, orthostatic tachycardia and OI symptoms.The subjects with POTS will be randomized, where TENS 7000 device will be placed to active and sham location.Autonomic symptoms assessment questionnaire (COMPASS-31),32 quality of life EQ-5D and neuropsychological tests
  Interventions: Diagnostic Test: Effect on inflammation after chronic PNS stimulation

INTERVENTIONS:
Diagnostic Test: Levels of inflammatory cytokine ( IL-6) in post-COVID-19 POTS and controls — Inflammatory and immune profile of post-COVID-19 POTS patients. Reduced PNS activity (vagal tone) in relation to persistent inflammation.
  Arms: Compare inflammatory markers (IL-6) in post- COVID 19 POTS patients with Controls
Diagnostic Test: Levels of inflammatory cytokine ( IL-6) in controls — Inflammatory and immune profile of healthy controls. Controls are the subjects who recovered from COVID-19 infection with no sequelae.
  Arms: Compare inflammatory markers (IL-6) in post- COVID 19 POTS patients with Controls
Diagnostic Test: Effect on inflammation after chronic PNS stimulation — Inflammatory biomarkers after restoring PNS function in post-COVID-19 POTS patients, by chronic transcutaneous vagus nerve stimulation (tVNS) in post COVID-19 POTS patients
  Arms: Effect of OI symptoms & inflmmation after Restoring PNS functions in post-COVID POTS patients.

SUMMARY:
The term post-acute COVID-19 syndrome or Long COVID is a disabling syndrome that persists beyond the 3-month convalescence period after COVID-19 infections.

This syndrome affects mostly women (~80%), present with chronic tachycardia and Orthostatic intolerance symptoms without any identifiable cause. In addition, non-specific symptoms such as fatigue, headache, and "brain fog", commonly described in POTS patients are also present in this novel condition, recently named post-COVID-19 tachycardia syndrome, POTS variant.

Reduced Vagal activity and unresolved inflammation is post-COVID-19 POTS is hypothesized as the cause of Long COVID

DETAILED DESCRIPTION:
Post-acute sequelae of COVID-19 infection or Long COVID is a growing concern, even in patients with mild initial illness. These patients develop numerous chronic debilitating symptoms including fatigue, chest pain, reduced exercise tolerance and tachycardia, with symptoms persisting weeks beyond the initial infection.

Preliminary data shows that post-COVID-19 POTS patients have reduced parasympathetic (PNS) function. Given that the PNS protects against inflammation, it is hypothesize that post-COVID-19 POTS is caused by reduced PNS activity, which in turn, contributes to persistent inflammation, orthostatic intolerance (OI) symptoms

Aim 1 of the study is to test the hypothesis that reduced PNS activity is associated with persistent inflammation in patients with post-COVID-19 POTS.

Aim 2: Test the hypothesis that restoring PNS function in post-COVID-19 POTS patients with chronic transcutaneous vagus nerve stimulation (tVNS) will improve inflammation, orthostatic tachycardia and OI symptoms.

Primary Outcome Measures:

1. To evaluate immune cell activation in post-COVID-19 POTS and patients with history of COVID-19 infection without sequelae and correlate this with the degree of decreased PNS activity. The primary endpoint is IL-6 levels.
2. Restoring PNS with chronic transcutaneous vagus nerve stimulation (tVNS), will improve the symptoms of orthostatic intolerance symptoms will

Rationale:

Elevated levels of IL-6, CRP and D-dimer are found in Long COVID patients, which resembles post-COVID tachycardia syndrome in POTS patients. Notably, stimulation of the efferent Vagus nerve has been shown to reduce cytokine production and systemic inflammation in response to endotoxin. Hence, decreased PNS function, as reported with acute SARS-CoV-2 infection and in post-COVID-19 POTS patients, may render these patients prone to persistent inflammation. The study aims to determine the link between PNS activity and immune activation in post-COVID-19 POTS.

Study population: Total of 60 participants, 30 post-COVID-19 POTS patients and 30 controls with history of COVID-19 infection without sequelae.

Study Visits: 5 visits, 3 in person and 1 telemedicine, Study procedures include EKG, urine and blood sample collection, Orthostatic Standing Test, Measurement of blood volume using carbon monoxide rebreathing technique, Tilt table test.

Participants will be asked to complete an autonomic symptoms assessment questionnaire (COMPASS-31),32 quality of life EQ-5D and neuropsychological tests that includes Cambridge Brain sciences: Web based cognitive assessment platform and PROMIS scale: Functional Activities Questionnaire in Older Adults with Dementia.

Transcutaneous Vagus Nerve Stimulation (tVNS): The device, which is FDA-approved TENS 7000 will be supplemented with ear clip electrodes, and the tragus or earlobe will be used as sites for vagal stimulation. The device will be used for 30 mins, twice a day for 28 days.

Randomization: The subjects will randomized to any one of the two sites of stimulation on the ear. There will be 50% chance to be allocated to one of the sites that may have less stimulation. The risk of having side effects is the same for both stimulation sites.

Data and Safety Monitoring Plan: The Data and Safety Monitoring Officer (DSMO) will provide objective review of treatment results as they relate to human safety and data quality. Dr. Cheryl Laffer, Professor of Medicine, Division of Clinical Pharmacology will serve as DSMO. The DSMO will review the initial protocol and will receive reports of the progress of the study every 12 months. These reports will provide information regarding recruiting, safety reporting, data quality, and efficacy.

Statistical Considerations:

Biostatistical Section Power analysis: The primary endpoint is serum IL-6. The proposed sample size of 60 (30 pairs of patients and controls) provides 90% power to detect an effect size of 0.62 for the mean difference in IL-6 between post-COVID-19 POTS (cases) and controls (COVID-19 infected w/o sequelae), with the two-sided type I error = 5%. This calculation is based on the preliminary data of mean difference of IL-6 ≈ 1.82 and the SD ≈ 2.94 in POTS.6 The effect size is defined as the ratio of mean IL-6 difference between cases and controls to standard deviation.

Data analysis plan: Demographic information will be tabulated. Descriptive statistics, including means, standard deviations, and ranges for continuous parameters, as well as percent and frequencies for categorical parameters, will be presented. T-test or Mann-Whitney (as appropriate) will be applied to examine the mean differences between cases and controls with respect to the outcomes. The conditional logistic regression model will be applied for the multivariable data analysis. The adjusted p-values and the adjusted 95% confidence intervals (CIs) will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Prior RT-PCR-confirmed COVID-19 infection.
* Post-COVID-19 POTS will be defined as the presence of orthostatic tachycardia (>30 bpm) and chronic (>3 months) pre-syncopal symptoms.

Exclusion criteria:

* Heart Disease: Myocardial Infarction, angina, heart failure
* History of stroke, or transient ischemic attack
* Undergone an invasive procedure for CVD (coronary artery bypass graft, angioplasty, valve replacement, pacemaker placement or other vascular surgeries)
* Uncontrolled hypertension defined as persistent blood pressure >140/90.
* Post-menopausal women.
* Diabetes Mellitus Type 1 or Type 2. ,
* Impaired Hepatic function
* Impaired renal function test (eGFR<60 mL/min/1.73m2).
* Ongoing substance abuse.
* Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study.
* History of seizures.
* Chronic use of steroids, NSAIDs.
* On biologics such as anti-IL6 (omalizumab) and anti-TNF-alpha drugs
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
IL-6 levels | Baseline to after 28 days of tVNS stimulation
  Evaluate immune cell activation in post-COVID-19 POTS and patients with history of COVID-19 infection without sequelae and correlate this with the degree of decreased PNS activity. The primary endpoint is IL-6 levels

SECONDARY OUTCOMES:
Orthostatic Symptoms Score | Baseline to after 28 days of tVNS stimulation
  Standardized Orthostatic Symptoms Score COMPASS-31: Composite Autonomic Symptom Score EQ-5D: as a Quality of Life Measure in People with Dementia AD8 Dementia Scale: The AD8 was developed as a brief instrument to help discriminate between signs of normal aging and mild dementia.
  E-cog test: Everyday Cognition scales (ECog) , an informant-rated questionnaire designed to detect cognitive and functional decline.

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, M.D, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States